CLINICAL TRIAL: NCT06641050
Title: External Validation of the TriAGE+ Score for Predicting Cerebrovascular Disease Risk in Patients Presenting With Dizziness in the Emergency Department
Brief Title: Validation of TriAGE+ for Predicting Stroke Risk in ED Patients Presenting With Dizziness
Status: Recruiting | Type: Observational
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emre Kudu, Principal Investigator, Marmara University Pendik Training and Research Hospital
Other Study IDs: 09.2024.240
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Stroke, Ischemic
Keywords: Triage+; Cerebrovascular Accident; Dizzyness; Neurologic Deficits
MeSH Terms: conditions — Ischemic Stroke; Stroke; Dizziness; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with dizziness: Individuals aged 18 years and over who present to the emergency department with dizziness will be assessed using the TriAGE+ score.
  Interventions: Diagnostic Test: Triage+ Score

INTERVENTIONS:
Diagnostic Test: Triage+ Score — The TriAGE+ score is used to evaluate the risk of cerebrovascular disease in patients presenting with dizziness. The score assists in determining the necessity of advanced diagnostic evaluation for stroke, potentially improving diagnostic accuracy and patient outcomes.

SUMMARY:
Ischemic cerebrovascular diseases originating from the brain's posterior circulation account for 20-25% of cases. Among patients diagnosed with cerebellar infarction, 10% present with isolated dizziness as their sole symptom. Notably, posterior circulation strokes and cerebellar infarcts are misdiagnosed 2 to 4 times more frequently than anterior circulation strokes. In 2017, Kuroda et al. developed the TriAGE+ score to assess stroke risk in patients presenting with dizziness. This study aims to externally validate the TriAGE+ score, focusing on its safety, applicability, and reliability in predicting cerebrovascular disease in the emergency department.

DETAILED DESCRIPTION:
Dizziness is a frequent complaint in emergency departments (ED), accounting for approximately 4% of visits. Epidemiological studies suggest that 3-20% of these patients experience dizziness due to cerebrovascular causes. In Turkey, data collected from 2013 to 2017 indicate that 2.4% of ED visits involved dizziness, with 36.8% of those patients being hospitalized due to central neurological events.

Cerebrovascular events (CVEs) involving the brain's posterior circulation-supplied by the vertebrobasilar arterial system and including regions such as the cerebellum, medulla oblongata, pons, and midbrain-are a common but often missed cause of dizziness. Studies have shown that 8.4% of patients presenting with isolated dizziness were later diagnosed with a posterior circulation stroke, and isolated dizziness has been recognized as the most common symptom in transient ischemic attacks (TIAs) and posterior circulation strokes.

In cerebellar stroke patients, 10% present with isolated dizziness. However, the National Institutes of Health Stroke Scale (NIHSS), which is commonly used to assess stroke severity, often underestimates posterior circulation strokes due to its focus on symptoms typically associated with anterior circulation infarcts. Posterior circulation strokes make up 20-25% of ischemic strokes, yet they are underdiagnosed 2 to 4 times more frequently than their anterior counterparts.

This diagnostic challenge underscores the need for an effective risk stratification tool to aid clinicians. Although several risk scores for cerebrovascular events exist, including the widely used ABCD2 score developed by Navi et al., they are often inadequate in assessing stroke risk in patients presenting with dizziness, as they emphasize unilateral weakness and speech impairment, both of which are less relevant to posterior circulation strokes.

In 2017, Kuroda et al. developed the TriAGE+ score to specifically predict stroke risk in patients presenting with dizziness. Their study, conducted in Japan across five emergency departments, included 498 patients. The score, which ranges from 0 to 17, was designed to categorize patients into four risk groups: low (<5), moderate (5-7), high (8-9), and very high (>9) risk for stroke. A threshold score of 10, determined through Receiver Operating Characteristic (ROC) analysis, provided a balance between sensitivity (77.5%; 95% CI 72.8-81.8) and specificity (72.1%; 95% CI 64.1-79.2). While this study demonstrated that the TriAGE+ score effectively predicted stroke risk, it was limited by its retrospective design and single-region focus, necessitating external validation.

Subsequently, Ho-Kun Yu et al. conducted an external validation study in Hong Kong in 2023, which, though supportive of the score's efficacy, shared similar limitations, including its retrospective, single-center design. As the TriAGE+ score was developed and validated primarily in Asia, it is critical to assess its generalizability and applicability in other populations. Our study seeks to perform an external validation of the TriAGE+ score in Turkey, with the aim of evaluating its safety, applicability, and reliability in a different population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dizziness who presented to the emergency department
* Patients who provide informed consent, or legal guardians providing consent for patients unable to do so.

Exclusion Criteria:

* Patients whose primary symptom is syncope or presyncope, or who present with dizziness due to hemodynamic compromise from gastrointestinal bleeding or other major events.
* Patients under the influence of alcohol or substances.
* Pregnant patients.
* Patients previously included in the study.
* Patients who refuse medical treatment or withdraw consent.
* Patients with incomplete data necessary for the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include adult (>18 years old) patients presenting to the emergency department with dizziness. These patients must provide informed consent, or consent must be obtained from their legal guardians if the patients are unable to do so. This population will serve as the basis for externally validating the TriAGE+ score, developed in Japan, in a Turkish emergency department setting.
Sampling Method: Non-Probability Sample
Enrollment: 841 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Stroke | 30 days (patient will be followed up 30 days based on their initial visit with dizziness. During the 30-day period, any subsequent visits to relevant specialities or the emergency department will be reviewed to assess for a stroke diagnosis.)
  The outcome for this study was the occurrence of stroke, defined as a new sudden neurological deficit of vascular origin.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No